CLINICAL TRIAL: NCT00154323
Title: A Multi-center, Randomized, Double-blind, Parallel Group, Placebo-controlled 52 Weeks Clinical Trial to Evaluate Efficacy and Safety of Oxcarbazepine p.o.(300-1200 mg/Day) as Adjuvant Therapy in the Bipolar Disorder I or II Treatment
Brief Title: The Efficacy and Safety of Oral Oxcarbazepine 300-1200 mg/Day as Adjuvant Therapy in the Treatment of Bipolar Disorder I or II This Study is Not Being Conducted in the United States.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CTRI476BES03
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Bipolar Disorder
Keywords: Oxcarbazepine, bipolar disorder
MeSH Terms: conditions — Bipolar Disorder | interventions — Oxcarbazepine

INTERVENTIONS:
Drug: Oxcarbazepine

SUMMARY:
Bipolar disorder is a psychiatric illness with clinical characteristics of mixed mania, grandiose delusions, and suicidality. This study will investigate the efficacy a safety of oxcarbazepine in the treatment of patients with bipolar disorder type I or II.

ELIGIBILITY:
Inclusion Criteria:

* History of bipolar disorder type I or II

Exclusion Criteria:

* Other serious medical conditions
* Treatment with antiepileptic medications

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2003-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Duration of remission

SECONDARY OUTCOMES:
Daily mood fluctuation
Time to new maniac/hypomanic episode
Time to new depressive episode
Number of relapsed patients at study completion and type/severity of episode
Change from baseline in functional activity

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Vieta, MD, Principal Investigator — Hospital Clinic, Universitary of Barcelona

REFERENCES:
- [Result] Vieta E, Cruz N, Garcia-Campayo J, de Arce R, Manuel Crespo J, Valles V, Perez-Blanco J, Roca E, Manuel Olivares J, Morinigo A, Fernandez-Villamor R, Comes M. A double-blind, randomized, placebo-controlled prophylaxis trial of oxcarbazepine as adjunctive treatment to lithium in the long-term treatment of bipolar I and II disorder. Int J Neuropsychopharmacol. 2008 Jun;11(4):445-52. doi: 10.1017/S1461145708008596. Epub 2008 Mar 17. PMID 18346292